CLINICAL TRIAL: NCT04487444
Title: A Pilot Trial of Thymalfasin (Ta1) to Treat COVID-19 Infection in Patients With Lymphocytopenia
Brief Title: Thymalfasin (Thymosin Alpha 1) to Treat COVID-19 Infection
Acronym: Ta1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to slow enrollment and the transfer of the PI to another institution.
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCN-16130571-2
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: thymosin alpha 1; lymphocytopenia; thymalfasin
MeSH Terms: conditions — COVID-19; Lymphopenia | interventions — Thymalfasin; Trace amine-associated receptor 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ta1 treatment arm (Experimental): Ta1 at a dose of 1.6 mg will be administered SC in 1 mL of diluent daily for a total of 1 week, in addition to standard of care.
  Interventions: Drug: Thymalfasin
- Control arm (No Intervention): No treatment will be provided in addition to standard of care.

INTERVENTIONS:
Drug: Thymalfasin — Synthetic 28 amino acid peptide identical to naturally circulating compound
  Other Names: Thymosin alpha 1; ZADAXIN (brand name); Ta1 (abbreviation)
  Arms: Ta1 treatment arm

SUMMARY:
It is our hypothesis that a course of Ta1 administered to hospitalized individuals with COVID-19 infection and lymphocytopenia will improve the time to recovery (primary objective) and severity of infection (secondary objectives) compared to untreated individuals in the same hospital with comparable lymphocytopenia.

After screening, hospitalized patients with COVID-19 and lymphocytopenia who meet the inclusion criteria will receive Ta1 (1.6 mg) administered subcutaneously (SC) daily for 1 week. Individuals in the control arm will be followed on the identical protocol but will not receive daily Ta1.

DETAILED DESCRIPTION:
Ta1 is a naturally occurring peptide that has been evaluated for its immunomodulatory activities and related therapeutic potential in several conditions and diseases, including infectious disease and cancer. ZADAXIN® brand Ta1 is a synthetic version currently approved for use in 37 countries; in particular it is approved in China for treatment of hepatitis B and to enhance vaccine response. Notably, Ta1 has been used clinically in pilot studies for treatment of severe acute respiratory syndrome (SARS) and other lung infections including acute respiratory distress syndrome (ARDS) and chronic obstructive pulmonary disorder (COPD), as well as infections after bone marrow transplant. Larger clinical trials have shown significant efficacy for treatment of severe sepsis and hepatitis B, along with certain cancers such as melanoma, hepatocellular, and lung cancer. Ta1 has also demonstrated improvement in response to vaccines in the elderly and in patients immunocompromised by renal disease.

Ta1 restores immune system homeostasis, by acting as multi-tasking protein depending on the host state of inflammation or immune dysfunction (such as infectious disease and cancer). Ta1 is believed to directly enhance the immune systems' recognition of infected cells and tumors cells, while also possibly modulating T cell activity and stimulating both innate and adaptive immunity to clear bacteria, virus, fungi and tumor cells. Ta1 serves a unique function in balancing pro-inflammatory and anti-inflammatory cytokine production through the regulation of distinct Toll-like receptors (TLRs) on different dendritic cell subsets. Data from other coronaviruses such as SARS-CoV and Middle Eastern respiratory syndrome (MERS)-CoV indicate that infection relies on their ability to impair both innate and adaptive immunity. During the 2003 pandemic, Ta1 was used as a prophylactic agent against SARS. Some published reports suggest that timely administration of immune-enhancers such as Ta1 to SARS patients was efficacious to a certain extent in controlling the development of the disease. Another study investigated the clinical manifestations, pharmacotherapy and prognosis of 46 patients with SARS and divided the severe cases (22 cases) into 2 groups according to administration of Ta1 and showed that the incidence rate of pulmonary fibrosis was lower in the group with Ta1 (2 of 14 cases) than the group without (6 out of 8 cases), i.e., 14.3% and 75.0%, respectively.

A recent study presented a retrospective analysis of hospitalized COVID-19 patients in China, in which those treated with Ta1 showed an improvement in lymphocyte subsets as well as a significant reduction in mortality (from 30 to 11%, p = 0.04).

Based on post-marketing treatment experience of more than 600,000 patients, Ta1 has been well tolerated. Ta1 has been administered to elderly subjects (up to 101 years old), children (as young as 13 months), and immunocompromised patients. The most common adverse events (AEs) in previous clinical trials include injection-site pain (such as burning and itching) which was mild and lasted for less than 30 minutes, as well as fever, nausea, and flu-like symptoms which were mild to moderate in severity. Thus, while Ta1 is one of only a few immunomodulatory agents that have been approved for human use, it does not appear to induce most of the side effects and toxicities commonly associated with other biological response modifiers (BRMs) in this class, such as interferon and interleukin (IL)-2.

The primary objective of the study is to determine whether Ta1 administered daily for one week to hospitalized COVID-19 patients with lymphocytopenia will improve time to recovery (free of respiratory failure) compared with a similar population of patients who do not receive Ta1. The secondary objectives are to determine whether hospitalized COVID-19 patients with lymphocytopenia treated with Ta1 will have a milder course of infection in terms of length of hospitalization stay, requirement (and length) for ICU stay, and requirement for supplemental oxygen or mechanical ventilation than patients not treated with Ta1, as well as higher chances of survival.

After screening, hospitalized patients with COVID-19 and lymphocytopenia who meet the inclusion criteria will receive Ta1 (1.6 mg) administered subcutaneously (SC) daily for 1 week. Individuals in the control arm will be followed on the identical protocol but will not receive daily Ta1. After the treatment period, all subjects will be followed and evaluated for efficacy outcomes at Day 14, with follow-up visits at Days 28, 42, and 60 (by phone, if the subject has been discharged from the hospital) to determine any AE/serious adverse event (SAE) and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* PCR positive for COVID-19 within the last 4 days
* Hospitalized
* SpO2 ≤ 93% on room air or requiring supplemental oxygen at screening (i.e. patients with severe disease)
* Lymphopenia (total lymphocyte count < 1.5 × 109/L)

Exclusion Criteria:

* Patients on mechanical ventilation
* Patients who are pregnant or breastfeeding
* Patients with multi-organ failure
* Patients with advanced malignancy receiving cytotoxic chemotherapy
* Patients with prior history of solid organ (kidney, liver, heart, lung, pancreas) or bone marrow transplant
* Patients on any other immunomodulatory therapy
* Patients receiving Plaquenil
* Patients who have participated in an investigational drug or device trial in previous 30 days
* Patients with a history of allergy or intolerance to Ta1
* Any other medical or psychiatric condition that, in the opinion of the Investigator, would compromise patient safety or interfere with the objectives of the protocol or completion of the protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Time to recovery (free of respiratory failure) | Day 28
  Length of time for patient to no longer require supplemental oxygen and can sustain a good oxygen saturation (SpO2) on room air

SECONDARY OUTCOMES:
Lymphopenia | Day 14
  Evaluation of CD4 and CD8 levels
Survival | Day 28
  Percentage of subjects still alive
Hospital length of stay | Day 28
  Length of time before hospital discharge
Requirement for high flow oxygen supplementation | Day 28
  Number of subjects that require high flow oxygen
Duration of high flow oxygen supplementation | Day 28
  Number of days that each subject requires high flow oxygen
ICU admission | Day 28
  Number of subjects that are admitted to the ICU
ICU length of stay | Day 28
  Number of days that each subject remains in the ICU
Mechanical ventilation | Day 28
  Number of subjects that require mechanical ventilation
Duration of mechanical ventilation | Day 28
  Number of days that each subject requires the mechanical ventilation
Change in any existing comorbidities (e.g., worsening congestive heart failure) or occurrence of newly diagnosed disease | Day 28
  Number of subjects that have decreases or increases in comorbidities existing at time of enrollment
Incidence of non-COVID-19 infections (other respiratory, urinary tract, cellulitis, etc.) | Day 28
  Number of subjects who get infections other than COVID-19
AEs/SAEs | Day 60
  Adverse events and serious adverse events experienced by the subjects
Changes to vital signs | Day 28
  Mild, moderate, or severe changes to vital signs (heart rate, blood pressure, temperature, number of respirations per minute) based on perceived clinical significance of the change
Changes in laboratory parameters | Day 28
  Mild, moderate, or severe changes to laboratory parameters (complete blood count and standard chemistry surveys) based on perceived clinical significance of the change

CONTACTS AND LOCATIONS:
Overall Officials: Eleftherios Mylonakis, MD PhD FIDSA, Principal Investigator — Lifespan
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu Y, Pan Y, Hu Z, Wu M, Wang C, Feng Z, Mao C, Tan Y, Liu Y, Chen L, Li M, Wang G, Yuan Z, Diao B, Wu Y, Chen Y. Thymosin Alpha 1 Reduces the Mortality of Severe Coronavirus Disease 2019 by Restoration of Lymphocytopenia and Reversion of Exhausted T Cells. Clin Infect Dis. 2020 Nov 19;71(16):2150-2157. doi: 10.1093/cid/ciaa630. PMID 32442287
- [Result] Shehadeh F, Benitez G, Mylona EK, Tran QL, Tsikala-Vafea M, Atalla E, Kaczynski M, Mylonakis E. A Pilot Trial of Thymalfasin (Thymosin-alpha-1) to Treat Hospitalized Patients With Hypoxemia and Lymphocytopenia Due to Coronavirus Disease 2019 Infection. J Infect Dis. 2023 Jan 11;227(2):226-235. doi: 10.1093/infdis/jiac362. PMID 36056913